CLINICAL TRIAL: NCT02856503
Title: Phase I/II Study Evaluating Safety and Effects of Preoperative High-Dose Vitamin D on the Receptors, Biomarkers and Pathological Characteristics of High Grade DCIS or Invasive Breast Cancer.
Brief Title: Effect of High Dose Vitamin D on Cancer Biomarkers and Breast Cancer Tumors
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: Eli Avisar (Other)
Responsible Party: Sponsor-Investigator, Eli Avisar, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20150288
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer; Invasive Breast Carcinoma; Ductal Carcinoma In-situ
Keywords: DCIS; IBC; Breast Cancer; Invasive Breast Carcinoma; High Grade Ductal Carcinoma in-situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1 - Group A - VD 3 Weeks (Experimental): Weekly oral dose of 50,000 IU Vitamin D3 (VD) for 3 weeks.
  Interventions: Drug: Vitamin D3
- Phase 1 - Group B - VD 4 Weeks (Active Comparator): Weekly oral dose of 50,000 IU Vitamin D3 (VD) for 4 weeks
  Interventions: Drug: Vitamin D3
- Phase 1 - Group C - VD 5 Weeks (Active Comparator): Weekly oral dose of 50,000 IU Vitamin D3 (VD) for 5 weeks.
  Interventions: Drug: Vitamin D3
- Phase 2 - VD (Experimental): Weekly oral dose of 50,000 IU Vitamin D3 (VD) therapy for the duration selected from the phase I part of the study.
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — Weekly oral dose of Vitamin D3 per protocol.
  Other Names: Toxiferol; Cholecalciferol

SUMMARY:
High-doses of Vitamin D (VD) may be used as targeted therapy against breast cancer. The investigators will assess the effect of high dose VD on the following biomarkers in the breast cancer cells: VDR, estrogen receptor (ER), progesterone receptor (PR), epidermal growth factor receptor 2 (Her2/neu), androgen receptor (AR), as well as epidermal growth factor receptor 1 (EGFR) and Ki-67, as markers of proliferation, and E-cadherin, a marker of invasion and metastasis.

DETAILED DESCRIPTION:
This is a phase I/II open-label, non-randomized study. In phase I, a fixed weekly course of oral high-dose Vitamin D (VD) is planned for either 3, 4 or 5 weeks; patients will be sequentially enrolled into 3 groups (A, B or C respectively) in a manner such that no more than two patients may have treatment-limiting toxicities (TLTs).

After the group with the optimal duration of VD therapy to achieve a "favorable response" is determined, phase II will begin enrollment.

Patients must be scheduled to have surgery performed within 2- weeks of the last dose of VD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed invasive breast carcinoma (IBC) or high grade (DIN3) Ductal Carcinoma in-situ (DCIS) and be scheduled for primary surgery.
2. Patients must be recommended/scheduled for primary surgery.
3. Female patients 18 years of age or older.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
5. Patients must have normal organ function as defined below:

   * Aspartate aminotransferase (AST/SGOT) < 4 times institutional upper limit of normal.
   * Alanine transaminase (ALT/SGPT) < 4 times institutional upper limit of normal.
   * Serum Bilirubin < 1.5 mg/dl.
   * Serum Alkaline Phosphatase < 4 times institutional upper limit.
   * Creatinine within normal institutional limits OR; Creatinine clearance >/= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.
   * Albumin within normal institutional limits
6. Women of childbearing potential (WoCBP) must have a negative (serum or urine) pregnancy test and agree to use barrier contraception while on treatment and for 30-days thereafter.
7. Ability to understand and the willingness to sign a written informed consent document by patient or their legal representatives.

Exclusion Criteria:

1. Previous history of breast cancer diagnosis or treatment.
2. Synchronous bilateral breast cancer.
3. Metastatic breast cancer
4. Patients recommended for neoadjuvant systemic therapy.
5. Patients may not be receiving any other investigational agents or have participated in any investigational drug study within 4 weeks preceding the start of study treatment.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with the study requirements.
7. Concurrent other malignancy
8. Uncontrolled hypertension
9. Chronic cholestatic or alcoholic liver disease
10. Chronic pancreatitis
11. Kidney impairment or renal stones
12. History of parathyroidectomy
13. Hypercalcemia, defined as serum level >11 mg/dl.
14. Abnormal laboratory data for: AST (SGOT), ALT (SGPT), Serum Bilirubin, Alkaline phosphatase, Creatinine and/or Creatinine clearance, and Albumin.
15. Patients receiving medications that are incompatible with VD.
16. Prior or known allergic reaction(s) to Vitamin D or other forms of Vitamin D.
17. Female patients who are pregnant or breast feeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1 - Rate of Treatment-Related Toxicity in Subjects | From Baseline to 30 days (+ 5 days) After Last Dose of Protocol Therapy, About 3 Months
  Rate of treatment-related adverse events and other toxicities in subjects.
Phase 2 - Rate of Favorable Treatment Response in Subjects Receiving Protocol Therapy Given Within the Optimal Duration Determined in Phase 1. | Up to 7 Weeks
  Rate of subjects achieving a "favorable treatment response" to protocol therapy given within the optimal duration determined in Phase 1. The effect of VD therapy will be assessed in terms of change in expression of VDR, ER, PR, HER2/neu, AR, Ki-67, E-cadherin and EGFR comparing surgical specimen (post-VD treatment) and baseline biopsy specimen (pre-VD treatment). The effect of VD will be described as increased expression, decreased expression or no change in expression of each marker/receptor measured.
  The expression of nuclear receptors/proteins (VDR, Ki-67, ER, PR, AR,) will be scored based on the percentage of positively staining nuclei as follows:
  * 0 (Negative) if <1%
  * +1 (Weak) if >1-10%
  * +2 (Moderate) if >10-50%
  * +3 (Strong) if >50%
  A decrease in the expression of Ki-67 by ≥+1 after treatment is considered a "favorable treatment response".

SECONDARY OUTCOMES:
Phase 1 - Optimal Duration of Once-Weekly Protocol Therapy | Up to 7 Weeks
  The determination of the optimal duration of once-weekly protocol therapy, 3, 4 or 5 weeks, as preoperative treatment to achieve a "favorable" treatment response in subjects with the study disease. The effect of VD therapy will be assessed in terms of change in expression of VDR, ER, PR, HER2/neu, AR, Ki-67, E-cadherin and EGFR comparing surgical specimen (post-VD treatment) and baseline biopsy specimen (pre-VD treatment). The effect of VD will be described as increased expression, decreased expression or no change in expression of each marker/receptor measured.
  The expression of nuclear receptors/proteins (VDR, Ki-67, ER, PR, AR,) will be scored based on the percentage of positively staining nuclei as follows:
  * 0 (Negative) if <1%
  * +1 (Weak) if >1-10%
  * +2 (Moderate) if >10-50%
  * +3 (Strong) if >50%
  A decrease in the expression of Ki-67 by ≥+1 after treatment is considered a "favorable treatment response".
Phase 2 - Rate of Treatment-Related Toxicity in Subjects | From Baseline to 30 days (+ 5 days) After Last Dose of Protocol Therapy, About 3 Months
  Rate of treatment-related adverse events and other toxicities in subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Eli Avisar, MD, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: No